CLINICAL TRIAL: NCT04549077
Title: Pulmonary Vascular Disease in Cystic Fibrosis
Brief Title: Pulmonary Vascular Disease in CF
Acronym: CF
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1239
Record Dates: First submitted 2020-08-09; First posted 2020-09-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Pulmonary Disease; Pediatric
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis Patients: Patients with Cystic Fibrosis.
- Historical Controls: Patients diagnosed with solid tumors, who have had a normal chest CT scan during screening for possible metastasis

SUMMARY:
In this project, the investigators seek to understand the role of endothelial cells in Cystic Fibrosis (CF) lung disease. This objective will be achieved by conducting a cross sectional clinical study to define the morphology of the pulmonary circulation across a range of lung function coupled with a mechanistic study of the effect of dysfunctional cystic fibrosis transmembrane conductance regulator (CFTR) in endothelial cells on vasculogenesis, epithelial morphogenesis and epithelial CFTR function. Toward that end, the investigators propose the following hypotheses; (a). Loss of pulmonary small blood vessels begins early in the CF lung and worsens with disease progression, (b).VEGFR2-CFTR interactions happen at the plasma membrane of endothelial cells and is likely to be involved in transendothelial ion transport (c) impaired VEGFR2-CFTR interactions on the endothelial cells will have a profound effect on vasculogenesis, epithelial morphogenesis and ion transport.

The first hypotheses will be tested through this clinical study. The following 2 hypotheses will be tested through laboratory studies that do not involve human subjects.

DETAILED DESCRIPTION:
Pulmonary disease in Cystic Fibrosis (CF) is characterized by progressive loss of functional gas exchange units that eventually results in respiratory failure. In CF lung disease, remodeling of pulmonary blood vessels, and vascular growth of bronchial blood vessels leading to systemic vascularization of the lung are the principal characteristics of pulmonary vascular disease. Studies have demonstrated that abnormal perfusion is present in up to 85% of 1 year old CF infants and only 17% of the perfusion deficits could be explained by mucus plugging or bronchial wall abnormalities at this age. Based on the investigators' state of the art method to reconstruct the pulmonary vasculature from non-contrast high resolution CT scan of the lungs, the investigators demonstrated that the blood volume in small vessels begins to decline when lung function is still in the normal range and worsens with increase disease severity. Furthermore, the investigators have also demonstrated that systemic vascularization of the lungs by the bronchial circulation begins at a FEV1% of 100. Preclinical studies of pulmonary endothelium revealed that delivering vascular endothelial growth factor receptor (VEGFR) antagonist to rats leads to air space enlargement and pruning of the pulmonary arterial tree. Thus, there is a central unanswered question as to whether pulmonary vascular disease (vascular remodeling and systemic vascularization) are just a squeal of parenchymal destruction or whether they contribute to the loss of alveolar gas exchange units and decline in lung function. In this proposal, the investigators will accomplish the following aims: 1) describe the morphology of the pulmonary vasculature across a wide range of lung function and relate the findings to functional outcomes, 2) examine mechanism of early loss of small blood vessels in CF patients as it relates to endothelial CFTR dysfunction. In addition, the investigators will study the changes in the pulmonary circulation after the initiation of triple combination therapy Trikafta (elexacaftor, ivacaftor, and tezacaftor).

This is a case control study of 93 cystic fibrosis patients and 100 age and gender matched controls. CF patients (cases) will be recruited from two cystic fibrosis centers, Cincinnati Children's Hospital and Riley Children's Hospital. Controls will be subjects from the oncology service without lung disease who had CT scan of the chest to rule out pulmonary metastasis. 31 subjects of the 93 subjects enrolled will receive a second evaluation 6 months after starting a clinically prescribed corrector / modulator of Cystic Fibrosis Transmembrane Conductance Protein Regulator (Trikafta) that was approved by the FDA in October, 2019 for patients with CF ages 12 and up. If FDA approval for use of Trikafta for ages 6-11 years of age is obtained, this patient age range will also be eligible for the second evaluation at 6 months.

ELIGIBILITY:
Cystic Fibrosis Patients:

Inclusion Criteria:

* 5-21 years of age
* diagnosis of CF based on a positive sweat test and genetic testing
* Baseline pulmonary condition defined as a) Absence of signs and symptoms of pulmonary exacerbation, b) Baseline pulmonary function test (PFT) defined as FEV1% that is no less than 5% of the best PFT in the previous 6 months, c) Patients should be off acute antibiotics for 2 weeks or longer.
* Subjects should be able to perform an acceptable and reproducible spirometry
* Study population will be equally divided between three groups based on FEV1%, (FEV1% ≥ 90); moderate (60 ≤ FEV1% < 90)

Exclusion Criteria:

* Enrollment in clinical trials of CFTR correctors and or potentiator
* Enrollment in gene therapy trial
* Pregnancy.

Historical Controls

Inclusion Criteria:

* solid tumor diagnosis
* had chest CT scan to survey possible metastasis or any other lung disease
* age and gender matched to Cystic Fibrosis patients

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 93 subjects with cystic fibrosis, 5-21 years of age, equally divided between males and females will be recruited from 2 CF centers; Cincinnati Children's Hospital and Riley Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The ratio (BV5/TBV) of blood volume in small < 5mm2 blood vessels (BV5) to the total pulmonary blood volume (TBV). | At baseline
  In Aim 1A, the reconstruction of pulmonary vasculature will be measured by the primary functional outcome variable, the ratio (BV5/TBV) of blood volume in small < 5mm2 blood vessels (BV5) to the total pulmonary blood volume (TBV).
The change in the the ratio (BV5/TBV) of blood volume in small < 5mm2 blood vessels (BV5) to the total pulmonary blood volume (TBV). | For a subset of 31 patients, the change in ratio will be measured between the baseline visit and 6 months post Trikafta therapy.
  In Aim 1A, the change in the reconstruction of pulmonary vasculature between the baseline and 6 month visit imaging will be measured by the primary functional outcome variable, the ratio (BV5/TBV) of blood volume in small < 5mm2 blood vessels (BV5) to the total pulmonary blood volume (TBV).

SECONDARY OUTCOMES:
Forced Expiratory Volume as a percent of the referenced value (FEV1%) | Baseline
  Forced Expiratory Volume as a percent of the referenced value (FEV1%)
The change in Forced Expiratory Volume as a percent of the referenced value (FEV1%) | For a subset of 31 patients, the change from baseline to 6 months post Trikafta therapy.
  The change in Forced Expiratory Volume as a percent of the referenced value (FEV1%)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No